CLINICAL TRIAL: NCT07027189
Title: DECIDE-AI:The Impact of Artificial Intelligence on Dentists' Decision-Making Process During Caries Detection: A Randomized Controlled Study
Brief Title: The Impact of Artificial Intelligence on Dentists' Decision-Making Process During Caries Detection
Acronym: DECIDE-AI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Prime Dental Alliance Eindhoven (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2025-18123
Record Dates: First submitted 2025-05-28; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Artificial Intelligence (AI) in Diagnosis; Artificial Intelligence Supported Image Reviewing
Keywords: Artificial Intelligence; Caries Detection; Decision-making; Dental Imaging; Treatment Planning
MeSH Terms: interventions — Artificial Intelligence; Diagnosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1: Caries detection without AI, Phase 2: Caries detection with AI (Active Comparator): In this group participants will examine caries lesions on the radiographs without AI support first. Then, after a wash-out period of one month, all participants will re-examine the same radiographs with AI.
  Interventions: Diagnostic Test: Artificial intelligence in diagnosis
- Phase 1: Caries detection with AI, Phase 2: Caries detection without AI (Active Comparator): In this group participants will examine caries lesions on the radiographs with AI support first. Then, after a wash-out period of one month, all participants will re-examine the same radiographs without AI.
  Interventions: Diagnostic Test: Artificial intelligence in diagnosis

INTERVENTIONS:
Diagnostic Test: Artificial intelligence in diagnosis — AI-based diagnostic programs have proved to enhance diagnostic performance, however research on its effects on treatment decisions is scarce. In contrast to other studies focusing on AI's accuracy or the resulting increase in dentists' accuracy, this study aims to investigate the differences in dentists' treatment recommendations when supported by AI versus when they are not during caries detection.

SUMMARY:
This study aims to evaluate the influence of artificial intelligence (AI) on the decision-making process for intervention after caries lesion detection. Participants will be dentists working in the Netherlands randomly divided into two groups. Dentists will be divided into two groups and receive a set of bitewing radiographs, which first will be evaluated with or without AI support according to their group. Participants will examine caries lesions on the radiographs and formulate treatment plans accordingly. Then, after a wash-out period of one month, the same radiographs, but in the opposite condition of AI support and again formulate treatment suggestions according to the present caries lesions.

DETAILED DESCRIPTION:
This crossover randomized controlled trial evaluates the effect of artificial intelligence (AI) decision support on dentists' treatment planning following caries detection bitewing radiographs. The study targets clinical decision-making processes by assessing how AI influences diagnostic interpretation and subsequent treatment suggestions. Dentists will be randomly assigned into two study arms. Each participant will evaluate a standardized set of digital bitewing radiographs under two conditions: once with AI assistance and once without, separated by a one-month wash-out period to minimize recall bias. The AI tool provides caries detection prompts based on radiographic analysis but does not suggest treatment. The crossover design enables within-subject comparison, controlling for individual diagnostic thresholds. The radiographs remain constant across both phases to isolate the influence of AI support. The study focuses on diagnostic performance and clinical decision outcomes, both with and without AI support. Treatment decisions are categorized into three predefined levels: no treatment, non-invasive treatment (e.g., fluoride application, polishing, sealing), and invasive intervention (i.e., restorative treatment). Diagnostic accuracy is measured against a reference standard and reported in terms of sensitivity and specificity. Caries detection will be classified using a modified International Caries Classification and Management System (ICCMS). This study design allows to quantify AI's impact on diagnostic performance, as well as on potential shifts in treatment approach. The study aims to contribute to evidence-based guidance on the integration of AI tools into clinical dental practice.

ELIGIBILITY:
Inclusion Criteria:

1. Graduated, practising dentists.
2. At least three years of experience

Exclusion Criteria:

1. Retired dentists.
2. Specialized practitioners (e.g., orthodontists and oral surgeons) if their typical practice does not involve routine caries diagnostics and treatment planning.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-02 (Estimated); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Treatment decisions: Compare the treatment recommendations of dentists for caries lesions detected with and without AI support. | Each participant will be assessed over a period of up to 2 months (includes both evaluation phases and washout period)
  The given options will be "no treatment", "non-invasive treatment" (fluoride varnish, polishing, sealing), and "restoration".
  Participants' answers will be compared to a reference standard.

SECONDARY OUTCOMES:
Diagnostic Accuracy in Caries Detection | Each participant will be assessed over a period of up to 2 months (includes both evaluation phases and washout period)
  RA0: No radiolucency - No visible caries. RA1: Radiolucency confined to the outer half of enamel - Enamel caries. RA2: Radiolucency extending to the inner half of enamel but not reaching dentin - Moderate enamel caries.
  RA3: Radiolucency extending into the outer third of dentin - Dentin caries. RA4: Radiolucency extending into the middle of dentin - Advanced dentin caries. RA5: Radiolucency extending into the inner third of dentin - Severe dentin caries.
  Participants' answers will be compared to a reference standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dentistry Radboud Uniersity Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Panyarak W, Wantanajittikul K, Suttapak W, Charuakkra A, Prapayasatok S. Feasibility of deep learning for dental caries classification in bitewing radiographs based on the ICCMS radiographic scoring system. Oral Surg Oral Med Oral Pathol Oral Radiol. 2023 Feb;135(2):272-281. doi: 10.1016/j.oooo.2022.06.012. Epub 2022 Jul 2. PMID 36513589
- [Background] Ayan E, Bayraktar Y, Celik C, Ayhan B. Dental student application of artificial intelligence technology in detecting proximal caries lesions. J Dent Educ. 2024 Apr;88(4):490-500. doi: 10.1002/jdd.13437. Epub 2024 Jan 10. PMID 38200405
- [Background] Mertens S, Krois J, Cantu AG, Arsiwala LT, Schwendicke F. Artificial intelligence for caries detection: Randomized trial. J Dent. 2021 Dec;115:103849. doi: 10.1016/j.jdent.2021.103849. Epub 2021 Oct 14. PMID 34656656
- [Background] Laske M, Opdam NJM, Bronkhorst EM, Braspenning JCC, van der Sanden WJM, Huysmans MCDNJM, Bruers JJ. Minimally Invasive Intervention for Primary Caries Lesions: Are Dentists Implementing This Concept? Caries Res. 2019;53(2):204-216. doi: 10.1159/000490626. Epub 2018 Aug 14. PMID 30107377
- [Background] Ammar N, Kuhnisch J. Diagnostic performance of artificial intelligence-aided caries detection on bitewing radiographs: a systematic review and meta-analysis. Jpn Dent Sci Rev. 2024 Dec;60:128-136. doi: 10.1016/j.jdsr.2024.02.001. Epub 2024 Feb 29. PMID 38450159
- [Background] Khanagar SB, Al-Ehaideb A, Maganur PC, Vishwanathaiah S, Patil S, Baeshen HA, Sarode SC, Bhandi S. Developments, application, and performance of artificial intelligence in dentistry - A systematic review. J Dent Sci. 2021 Jan;16(1):508-522. doi: 10.1016/j.jds.2020.06.019. Epub 2020 Jun 30. PMID 33384840
- See also: Dutch professional profile description for dentists. — https://knmt.nl/sites/default/files/platform/20211220_functieprofiel_tandarts.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT07027189/Prot_SAP_000.pdf